CLINICAL TRIAL: NCT07380945
Title: Development of A Multi-section Olfactory Cleft Opacity Staging System in Patients With Central Compartment Atopic Disease (CCAD)
Brief Title: Development of A Multi-section Olfactory Cleft Opacity Staging System in Patients With CCAD
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Dawei Wu, Associate Researcher, Peking University Third Hospital
Other Study IDs: 9059105
Record Dates: First submitted 2026-01-24; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Central Compartment Atopic Disease (CCAD)
Keywords: olfactory cleft; olfactory dysfuction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with CCAD
  Interventions: Other: Computer Tomography
- non-CCAD patients with chronic rhinosinusitis
  Interventions: Other: Computer Tomography

INTERVENTIONS:
Other: Computer Tomography — low-dose CT is taken
  Other Names: collection of the percentage of peripheral blood eosinophils

SUMMARY:
This study aims to develop a modified CT scoring system to evaluate the association between olfactory cleft obstruction patterns and olfactory dysfunction in patients with central region atopic disease (CCAD).

The main questions that the clinical trial aims to answer are: Can this modified CT scoring system be used to assess the degree of olfactory impairment in patients with CCAD? How well does the modified CT score correlate with the patient's olfaction compared to the traditional CT score?

DETAILED DESCRIPTION:
Olfactory dysfunction is one of the important clinical manifestations of patients with central compartment atopic disease (CCAD), whose pathological mechanism has not been fully elucidated. Previous studies have shown that physical blockage of Olfactory Cleft (OC) may block odor molecules from reaching the olfactory mucosa in the olfactory region.

At present, there is still a lack of systematic standards for imaging evaluation of olfactory obstruction patterns. Traditional CT scores are mostly based on the percentage of occlusion area in a single dimension, which is difficult to reflect the turbidity of the anterior and posterior OC. The anterior olfactory cleft serves as the main entrance to the odor molecules, and its apical and middle lower blockage may have different effects on olfactory conduction. Therefore, it is urgent to establish a regionally divided CT scoring system to more accurately analyze the spatial characteristics of olfactory cleft opacification in CCAD patients and its correlation with olfactory function.

This prospective study aims to develop an improved olfactory CT scores evaluation system to reveal the anatomical mechanism of olfactory dysfunction in patients with CCAD. All the participants (n=??) had undergone:

1. Clinical assessment of olfactory function Using the Sniffin' Sticks Test to evaluate olfaction. The scores of the three tests of odor threshold (OT), odor discrimination (OD) and odor identification (OI) are added to the total TDI score. TDI with a total score of 48 points is normal for people >30.75 points, ≤30.75 is classified as olfactory disorder, among which 16-30 indicates hyposmia and <16 indicates anosmia. Patients are divided into three groups according to the TDI score.
2. Traditional CT scores The olfactory cleft was considered to start at the anterior most olfactory filament (the anterior plane of middle turbinate) and end just anterior to the face of the sphenoid sinus. A computed tomography (CT) scan was performed to evaluate the OC opacification. The anterior end of the superior turbinate is boundary, and the OC is divided into two parts: anterior and posterior. The OC opacifications, in which the normal airway filled with a value representing soft tissue and /or presence of close contact between the nasal turbinates and the nasal septum, were graded on a scale of 0-4 by the ratio of the opacified area to the whole area of the corresponding region of the olfactory cleft, with 0 (no opacification), 1 (25%), 2 (25%-50%), 3 (50%-75%), and 4 (>75%).
3. Modified olfactory cleft scores The scores of the independently assessed regions including the left anterior, left posterior, right anterior, and right posterior olfactory cleft are summed to obtain the anterior (left anterior and right anterior), posterior (left posterior and right posterior) , and total scores. Specifically, the opacification of each OC subregion is independently assessed, with a score of 1 if unilateral opacity is observed, 2 points for bilateral opacity, and 0 if none.

ELIGIBILITY:
Inclusion Criteria for patient group:

1. Diagnosed with CCAD based on the diagnostic criteria of the EPOS guideline.
2. Provision of signed and dated informed consent form.

Inclusion Criteria for control group:

1. Diagnosed with CRS (non-CCAD) based on the diagnostic criteria of the EPOS guideline.
2. Provision of signed and dated informed consent form.

Exclusion Criteria for patient group:

1. Those who have taken oral glucocorticoids, antibiotics, anti-leukotrienes, and antihistamines within four weeks.
2. Patients who have had prior sinus surgery.
3. Patients with fungal sinusitis, inverted papilloma, or other nasal diseases.
4. Patients with a diagnosis of immune suppression or suspicion of malignancy that may be affecting the nose/paranasal sinuses.
5. Patients who are mentally or physically unable to perform olfactory tests

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients were recruited from the Department of Otolaryngology at Peking University Third Hospital in clinic.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the novel olfactory cleft CT scoring system for imaging assessment in CCAD patients | Immediately after CT scans
  Validation of the novel CT scoring system for superior characterization of olfactory cleft obstruction compared to the traditional CT scoring system.
Predictive performance of the novel olfactory cleft CT scoring system | Immediately after CT scans
  Construct a predictive model for CCAD using logistic regression, incorporating both the novel CT score and peripheral blood eosinophil percentage, and compare it with the traditional olfactory cleft CT scoring system.

SECONDARY OUTCOMES:
Correlation between novel olfactory cleft CT scores in different regions and CCAD diagnosis | Immediately after CT scans
  Analyze the differences in scoring across various anatomical subregions in the CCAD group and identify the most diagnostically relevant regions.
Association between the novel olfactory cleft CT score, olfactory function, and eosinophil percentage | Immediately after CT scans
  Investigate the relationship between the novel CT scoring system and olfactory dysfunction, as well as its potential to reflect Type 2 inflammation (eosinophilic activity).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Otolaryngology Head and Neck Surgery, Peking University Third Hospital, Beijing, People's Republic of China, China

IPD SHARING:
Plan to Share IPD: No
We will decide whether to share the individual participant data after the study.